CLINICAL TRIAL: NCT05099159
Title: A Double-blind, Randomized, Placebo-controlled Multicenter Study to Investigate Efficacy and Safety of Elinzanetant for the Treatment of Vasomotor Symptoms Over 26 Weeks in Postmenopausal Women
Brief Title: A Study to Learn More About How Well Elinzanetant Works and How Safe it is for the Treatment of Vasomotor Symptoms (Hot Flashes) That Are Caused by Hormonal Changes Over 26 Weeks in Women Who Have Been Through the Menopause (OASIS-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21652; 2020-004855-34 (EudraCT Number)
Record Dates: First submitted 2021-10-19; First posted 2021-10-29 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Vasomotor Symptoms Associated With Menopause; Hot Flashes
Keywords: Menopause
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elinzanetant (BAY3427080) (Experimental): Participants will receive 120 mg elinzanetant orally once daily for 26 weeks.
  Interventions: Drug: Elinzanetant (BAY3427080)
- Placebo + elinzanetant (Placebo Comparator): Participants will receive matching placebo orally once daily for 12 weeks, followed by elinzanetant 120 mg for 14 weeks.
  Interventions: Drug: Elinzanetant (BAY3427080); Drug: Placebo

INTERVENTIONS:
Drug: Elinzanetant (BAY3427080) — 120 mg elinzanetant orally once daily
Drug: Placebo — Matching placebo orally once daily
  Arms: Placebo + elinzanetant

SUMMARY:
Researchers are looking for a better way to treat women who have hot flashes after women have been through the menopause. Hot flashes are caused by the hormonal changes that happen when a woman's body has been through the menopause. Menopause is when women stop having a menstrual cycle, also called a period. During the menopause, the ovaries increasingly produce less sex hormones as a result of the natural ageing process and related hormonal adjustments. The decline in hormone production can lead to various symptoms which, in some cases, can have a very adverse effect on a menopausal woman's quality of life.

The study treatment, elinzanetant, was developed to treat symptoms caused by hormonal changes. It works by blocking a protein called neurokinin from sending signals to other parts of the body, which is thought to play a role in starting hot flashes. There are treatments for hot flashes in women who have been through the menopause, but may cause medical problems for some people.

In this study, the researchers will learn how well elinzanetant works compared to a placebo in women who have been through the menopause and have hot flashes. A placebo looks like a treatment but does not have any medicine in it. To compare these study treatments, the doctors will ask the participants to record information about the participants' hot flashes in an electronic diary. The researchers will study the number of hot flashes the participants have and how severe the hot flashes are. The researchers will look at the results from before treatment, after 4 weeks, and after 12 weeks of treatment.

The participants in this study will take two capsules of either elinzanetant or the placebo once a day. The participants who take elinzanetant will take it for 26 weeks. The participants who take the placebo will take it for 12 weeks and then take elinzanetant for the next 14 weeks.

During the study, the participants will visit the site approximately 9 times and perform 1 visit by phone. Each participant will be in the study for approximately 36 weeks. The treatment duration will be 26 weeks.

During the study, the participants will:

* record information about the participants' hot flashes in an electronic diary
* answer questions about the participants' symptoms

The doctors will:

* check the participants' health
* take blood samples
* ask the participants questions about what medicines the participants are taking and if the participants are having adverse events An adverse event is any medical problem that a participant has during a study. Doctors keep track of all adverse events that happen in studies, even if doctors do not think the adverse events might be related to the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal, defined as:

  1. at least 12 months of spontaneous amenorrhea prior to signing of informed consent, or
  2. at least 6 months of spontaneous amenorrhea prior to signing of informed consent with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL and a serum estradiol concentration of < 30 pg/mL, or
  3. at least 6 months after hysterectomy at signing of informed consent with serum FSH levels > 40 mIU/mL and a serum estradiol concentration of < 30 pg/mL, or
  4. surgical bilateral oophorectomy with or without hysterectomy at least 6 weeks prior to signing of informed consent.
* Moderate to severe hot flash (HF) associated with the menopause and seeking treatment for this condition.
* Participant has completed Hot Flash Daily Diary (HFDD) for at least 11 days during the two weeks preceding baseline visit, and participant has recorded at least 50 moderate or severe HF (including night-time HF) over the last 7 days that the HFDD was completed (assessed at the Baseline Visit).

Exclusion Criteria:

* Any clinically significant prior or ongoing history of arrhythmias, heart block and QT prolongation either determined through clinical history or on ECG evaluation.
* Any active ongoing condition that could cause difficulty in interpreting vasomotor symptoms (VMS) such as: infection that could cause pyrexia, pheochromocytoma, carcinoid syndrome.
* Current or history (except complete remission for 5 years or more) of any malignancy (except basal and squamous cell skin tumors). Women receiving adjuvant endocrine therapy (e.g. tamoxifen, aromatase inhibitors, GnRH analogues) cannot be enrolled in this study.
* Uncontrolled or treatment-resistant hypertension. Women with mild hypertension can be included in the study if they are medically cleared prior to study participation.
* Untreated hyperthyroidism or hypothyroidism.

  * Treated hyperthyroidism with no abnormal increase of thyroid function laboratory parameters and no relevant clinical signs for > 6 months before signing of informed consent is acceptable.
  * Treated hypothyroidism with normal thyroid function test results during screening and a stable (for ≥ 3 months before signing of informed consent) dose of replacement therapy is acceptable.
* Any unexplained post-menopausal uterine bleeding.
* Clinically relevant abnormal findings on mammogram.
* Abnormal liver parameters.
* Disordered proliferative endometrium, endometrial hyperplasia, polyp, or endometrial cancer diagnosed based on endometrial biopsy during screening.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2021-10-29 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-10-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (113):
- United States (48):
  - Accel Research Sites | Cahaba Medical Care - Birmingham, AL, Birmingham, Alabama
  - Women's Health Alliance of Mobile, Mobile, Alabama
  - Onyx Clinical Research - Peoria, Peoria, Arizona
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - National Institute of Clinical Research - Garden Grove, Garden Grove, California
  - Clinical Trials Research - Lincoln, Lincoln, California
  - Torrance Clinical Research Institute, Inc. | Lomita, CA, Lomita, California
  - Women's Health Care Research | San Diego, CA, San Diego, California
  - Advanced Women's Health Institute | Denver Office, Greenwood Village, CO, Greenwood Village, Colorado
  - Physicians' Research Options, LLC | Red Rocks OBGYN, Lakewood, Colorado
  - Helix Biomedics, LLC, Boynton Beach, Florida
  - Clinical Research of West Florida | Clearwater, FL, Clearwater, Florida
  - Sweet Hope Research Specialty, Inc. - Miami Lakes, Hialeah, Florida
  - Ocean Blue Medical Research Center, Inc | Miami Springs, FL, Miami Springs, Florida
  - Suncoast Clinical Research Inc. | Pasco, New Port Richey, Florida
  - Sensible Healthcare, LLC, Ocoee, Florida
  - Clinical Research of West Florida | Tampa, FL, Tampa, Florida
  - Fellows Research Alliance, Inc | Savannah, GA, Savannah, Georgia
  - Family Care Research | Boise, ID, Boise, Idaho
  - Leavitt Clinical Research | Idaho Falls, ID, Idaho Falls, Idaho
  - University of Chicago | Laboratory of Dr. Al-Hendy, Chicago, Illinois
  - AMR - Chicago, Oak Brook, Illinois
  - Clinical Trials Management | Northshore Office, Covington, Louisiana
  - Tandem Clinical Research | Marrero, LA, Marrero, Louisiana
  - Ob and Gyn Physicians MidAtlantic - SKYCRNG, Oxon Hill, Maryland
  - Genesis Clinical Research and Consulting, LLC, Fall River, Massachusetts
  - Saginaw Valley Medical Research Group, LLC | Saginaw, MI, Saginaw, Michigan
  - Metro Jackson OBGYN | Jackson, MS, Jackson, Mississippi
  - R. Garn Mabey Jr. M.D. Gynecology, Las Vegas, Nevada
  - Capital Health | Capital Health OBGYN Lawrenceville, Lawrenceville, New Jersey
  - Columbia University Medical Center, New York, New York
  - Eastern Carolina Women's Center | New Bern, NC, New Bern, North Carolina
  - Unified Women's Clinical Research | Raleigh, NC, Raleigh, North Carolina
  - OHSU Hospital - OB-GYN - Women's Health Research Unit, Portland, Oregon
  - UPMC Magee-Women's Hospital - Gynecology, Pittsburgh, Pennsylvania
  - Tribe clinical Research LLC | Greenville, SC, Greenville, South Carolina
  - Medical Research Center of Memphis | Memphis, TN, Memphis, Tennessee
  - Research Memphis Associates, LLC | Memphis, TN, Memphis, Tennessee
  - Austin Regional Clinic | ARC Kelly Lane, Austin, Texas
  - DiscoveResearch, Inc., Bryan, Texas
  - South Texas Clinical Research, Corpus Christi, Texas
  - Sig Gyn Services (Dr. John A. Whitfield, MD) | Fort Worth, TX, Fort Worth, Texas
  - Advances in Health, INC. | Houston, TX, Houston, Texas
  - UTHealth Womens Research Program | Memorial City, Houston, Texas
  - ClinRx Research, LLC, Plano, Texas
  - The Woman's Place - Midlife Health, Charlottesville, Virginia
  - Tidewater Clinical Research, Inc., Norfolk, Virginia
  - Northwest Clinical Research Center | Bellevue, WA, Bellevue, Washington
- Canada (10):
  - Alta Clinical Research Inc | Edmonton, Canada, Edmonton, Alberta
  - IWK Health Centre | Department of Obstetrics and Gynaecology, Halifax, Nova Scotia
  - Ecogene 21, Chicoutimi, Quebec
  - GCP Research | Montreal, Canada, Montreal, Quebec
  - Clinique Ovo | R&D Department, Montreal, Quebec
  - Diex Recherche Sherbrooke Inc., Sherbrooke, Quebec
  - Alpha Recherche Clinique | Val-Belair, Val-Bélair, Quebec
  - Diex Recherche Victoriaville Inc., Victoriaville, Quebec
  - Diex Recherche Quebec Inc., Québec
  - Alpha Recherche Clinique | Lebourgneuf, Québec
- Czechia (5):
  - GynPorCentrum s.r.o., Krnov
  - MUDr. Martina Maresova Rosenbergova, gynekologie, Pilsen
  - Gynekologie Studentsky dum s.r.o., Prague
  - GYNEVI s.r.o., Rokycany
  - Gynpraxetabor s.r.o., Tábor
- Germany (10):
  - Synexus Frankfurt Clinical Research Centre, Frankfurt am Main, Hesse
  - Praxis Hr. Dr. S. Fiedler, Aachen, North Rhine-Westphalia
  - Frauenärzte am Schloss Borbeck, Essen, North Rhine-Westphalia
  - Medplus Nordrhein, Krefeld, North Rhine-Westphalia
  - Synexus Leipzig Clinical Research Centre, Leipzig, Saxony
  - Praxis f. Gynäkologie und Geburtshilfe, Bernburg, Saxony-Anhalt
  - Frauenarztpraxis Dr. Inka Kiesche, Halle, Saxony-Anhalt
  - Femme Frauenarztpraxis, Gera, Thuringia
  - emovis GmbH, Berlin
  - Synexus Berlin Clinical Research Centre, Berlin
- Italy (4):
  - A.O.U. Policlinico Federico II Napoli, Naples, Campania
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Azienda Ospedaliera Ordine Mauriziano Di Torino, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Integrata Verona_Borgo Trento - Ostetricia e Ginecologia B, Verona, Veneto
- Norway (5):
  - Kirkeparken Spesialistpraksis, Fredrikstad
  - Medicus | Oslo, Norway, Oslo
  - Oslo University Hospital | Division of Obstetrics and Gynecology, Department of Research, Oslo
  - Medicus | Stavanger, Norway, Stavanger
  - Medicus AS, Trondheim
- Poland (6):
  - Gabinet Ginekologiczny Janusz Tomaszewski, Bialystok
  - CLINICAL MEDICAL RESEARCH Sp. z o. o., Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Vita Longa Sp. z o.o., Katowice
  - Etyka Osrodek Badan Klinicznych, Olsztyn
  - Twoja Przychodnia - Szczecinskie Centrum Medyczne, Szczecin
- Portugal (7):
  - Luz Saude | Hospital Beatriz Angelo - Centro de Investigacao Clinica, Loures, Lisbon District
  - Hospital Santa Maria | Centro de Investigacao Clinica, Missing, Lisbon District
  - Hospital Pedro Hispano | Clinical Research Center, Matosinhos Municipality, Porto District
  - Luz Saude | Hospital da Luz Setubal - Clinical Research Department, Setúbal, Setúbal District
  - Centro Hospitalar e Universitario de Coimbra, E.P.E. | Department of Gynecology, Coimbra
  - Centro Hospitalar de Lisboa Ocidental | Clinical Research Department, Lisbon
  - Centro Hospitalar Universitario do Porto | Servico de Investigacao Clinica, Porto
- RC Medical, Novosibirsk, Russia
- Slovakia (6):
  - Univerzitna nemocnica Bratislava, Nem. Sv. Cyrila a Metoda, Bratislava
  - GYNARIN, s.r.o., Fiľakovo
  - ULMUS, s r.o., Hlohovec
  - Nemocnica AGEL Kocice-Saca a.s., Kosice - Saca
  - GA Lucenec s.r.o, Lučenec
  - Virina sano, s.r.o. Gynekologicko porodnicka ambulancia, Veľký Krtíš
- Switzerland (5):
  - Kantonsspital Baden, Baden, Canton of Aargau
  - Universitätsspital Basel, Basel, Canton of Basel-City
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Inselspital Universitätsspital Bern, Bern
  - UniversitätsSpital Zürich, Zurich
- Ukraine (6):
  - Ivano-Frankivsk Regional Perinatal Center, Ivano-Frankivsk
  - Instr. of Pediatrics, Obstetrics & Gynecology, Kiev
  - Center of innovative medical technologies of NAS of Ukraine, Kiev
  - Medical Center LLC "Verum Expert Clinic", Kyiv
  - Medical Center Motor Sich, Zaporizhzhya
  - CNE "Zaporizhzhia Regional Clinical Hospital" of Zaporizhzhia regional council, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- [Derived] Pinkerton JV, Simon JA, Joffe H, Maki PM, Nappi RE, Panay N, Soares CN, Thurston RC, Caetano C, Haberland C, Haseli Mashhadi N, Krahn U, Mellinger U, Parke S, Seitz C, Zuurman L. Elinzanetant for the Treatment of Vasomotor Symptoms Associated With Menopause: OASIS 1 and 2 Randomized Clinical Trials. JAMA. 2024 Aug 22;332(16):1343-54. doi: 10.1001/jama.2024.14618. Online ahead of print. PMID 39172446
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=21652&attachmentIdentifier=360af6f8-5cb7-4bf8-9165-138cb3fcb475&fileName=21652_Study_Synopsis_CTP.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217261&parentIdentifier=21652&attachmentIdentifier=7382b90d-9960-4a5e-9866-8df8ff0fc974&fileName=21652_PLS_Final_Clean_copy_08Oct2024.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 95 study centers in 10 countries worldwide, between 29-Oct-2021 (first participant first visit) and 10-Oct-2023 (last participant last visit).
Pre-assignment Details: A total of 1483 participants were screened, of whom 1083 participants were screen failures. Most common reason for screen failure was not meeting the eligibility criteria (1044 participants). 400 of the screened participants were randomized to treatment and 324 participants completed the study.
Groups:
- Elinzanetant 120 mg: Participants received elinzanetant 120 mg orally once daily for 26 weeks
- Placebo - Elinzanetant 120 mg: Participants received placebo for 12 weeks, followed by elinzanetant 120 mg orally once daily for 14 weeks
Period: Overall Study
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Started | 200 | 200
Completed | 157 | 167
Not Completed | 43 | 33
Not completed — Subject Decision | 14 | 10
Not completed — Adverse Event | 7 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Lost to Follow-up | 6 | 1
Not completed — Non-compliance with study drug | 1 | 4
Not completed — Other | 1 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Did not complete study treatment but completed FU | 13 | 12

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was analyzed. FAS: all randomized subjects were included. Subjects in the full analysis set were analyzed according to the randomized intervention (intention-to-treat).
Groups:
- Total: Total of all reporting groups
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (5.0) | 54.4 (4.5) | 54.6 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 200 | 200 | 400
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 24 | 37
  Not Hispanic or Latino | 186 | 175 | 361
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 25 | 60
  White | 163 | 172 | 335
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 4 (Assessed by HFDD)
Description: Participants' assessments of HF were recorded electronically twice daily using the sponsor developed Hot Flash Daily Diary (HFDD). The HFDD was completed in the morning after waking up (morning diary) and each evening at bedtime (evening diary) on the hand-held device. The HFDD items assessed the number of mild, moderate, and severe HF experienced during the day and during the night. Mild HF was defined as a "sensation of heat without sweating", moderate HF was defined as a "sensation of heat with sweating, but able to continue activity", and severe HF was defined as a "sensation of heat with sweating, causing cessation (stopping) of activity".
  The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically, for Week 4, Day 22-28 were used (Day 1 corresponds to start of treatment).
Time Frame: From baseline to Week 4
Population: FAS
Measure: Mean (Standard Deviation); unit: Hot Flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Hot Flashes per day
  Baseline: number analyzed (Participants) | 199 | 200
  Baseline | 14.66 (11.08) | 16.16 (11.15)
  Change from Baseline: number analyzed (Participants) | 185 | 192
  Change from Baseline | -8.58 (9.16) | -6.07 (8.91)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, Mixed model repeated measures (MMRM) — One-sided. A multiplicity adjustment strategy was defined using the graphical approach, controlling the overall type I error rate at a one-sided alpha level of 0.025 for confirmatory statistical superiority testing; Least squares (LS) means = -3.04, 95% CI 2-sided [-4.40 to -1.68]

2. Primary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 12 (Assessed by HFDD)
Description: The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically, for Week 12, Day 78-84 were used (Day 1 corresponds to start of treatment).
Time Frame: From baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Hot flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Hot flashes per day
  Baseline: number analyzed (Participants) | 199 | 200
  Baseline | 14.66 (11.08) | 16.16 (11.15)
  Change from Baseline: number analyzed (Participants) | 174 | 180
  Change from Baseline | -9.96 (10.25) | -7.24 (8.49)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; LS-means = -3.24, 95% CI 2-sided [-4.60 to -1.88]

3. Primary Outcome: Mean Change in Severity of Moderate to Severe HF From Baseline to Week 4 (Assessed by HFDD)
Description: In the HFDD, hot flash (HF) severity is scored as 1=mild, 2=moderate, and 3=severe; a decrease indicates improvement. The diary records the number of mild, moderate, and severe HFs during day and night. Mild HFs are a "sensation of heat without sweating"; moderate are "heat with sweating but able to continue activity"; severe are "heat with sweating that stops activity."
  Baseline mean daily severity is calculated as:
  (2×moderateHFs+3×severeHFs)÷(totalmoderate+severeHFs).(2 × moderate HFs + 3 × severe HFs) ÷ (total moderate + severe HFs).(2×moderateHFs+3×severeHFs)÷(totalmoderate+severeHFs).
  If none occur, severity=0. Weekly severity during treatment is based on available days (Week 4: Days 22-28; Week 12: Days 78-84; Day 1=start of treatment), averaging the mean daily severity for that week. If more than 2 days are missing, the weekly value is set to missing
Time Frame: From baseline to Week 4
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Units on a scale
  Baseline: number analyzed (Participants) | 199 | 200
  Baseline | 2.53 (0.24) | 2.54 (0.24)
  Change from Baseline: number analyzed (Participants) | 185 | 192
  Change from Baseline | -0.75 (0.68) | -0.53 (0.55)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p = 0.0003, MMRM — [p-value comment as in outcome 1, analysis 1]; LS-means = -0.22, 95% CI 2-sided [-0.34 to -0.09]

4. Primary Outcome: Mean Change in Severity of Moderate to Severe HF From Baseline to Week 12 (Assessed by HFDD)
Description: In the HFDD, hot flash (HF) severity is categorized as 1=mild, 2=moderate, 3=severe; thus, a decrease indicates improvement. The HFDD records the number of mild, moderate, and severe HFs during day and night. Mild HFs are a "sensation of heat without sweating"; moderate involve "heat with sweating but able to continue activity"; severe involve "heat with sweating that stops activity."
  Mean daily severity at baseline is calculated as:
  (2 × moderate HFs) + (3 × severe HFs)] ÷ (total moderate + severe HFs). If none occur, severity is set to 0. Weekly severity during treatment is based on available days (Week 4: Days 22-28; Week 12: Days 78-84; Day 1=start of treatment), averaging mean daily severity across that week. If more than 2 days are missing, the week is set to missing.
Time Frame: From baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Units on a scale
  Baseline: number analyzed (Participants) | 199 | 200
  Baseline | 2.53 (0.24) | 2.54 (0.24)
  Change from baseline: number analyzed (Participants) | 174 | 180
  Change from baseline | -0.97 (0.78) | -0.65 (0.67)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; LS-means = -0.29, 95% CI 2-sided [-0.44 to -0.14]

5. Secondary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline to Week 1 (Assessed by HFDD)
Description: Participants' assessments of HF were recorded electronically twice daily using the sponsor developed HFDD. The HFDD was completed in the morning after waking up (morning diary) and each evening at bedtime (evening diary) on the hand-held device.
Time Frame: From baseline to Week 1
Population: FAS
Measure: Mean (Standard Deviation); unit: Hot flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Hot flashes per day
  Baseline: number analyzed (Participants) | 199 | 200
  Baseline | 14.66 (11.08) | 16.16 (11.15)
  Change from baseline: number analyzed (Participants) | 198 | 197
  Change from baseline | -4.66 (6.70) | -3.57 (6.86)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p = 0.0013, MMRM — [p-value comment as in outcome 1, analysis 1]; LS-means = -1.66, 95% CI 2-sided [-2.73 to -0.58]

6. Secondary Outcome: Mean Change in Frequency of Moderate to Severe HF From Baseline Over Time (Assessed by HFDD)
Description: The frequency of moderate to severe HF for each week during the treatment period was calculated using the available data during that particular week. Specifically, for Week 1 Days 2-8 were used instead of 1-7, because the intake started on Day 1 only before going to bed, for Week 4 Days 22-28 were used and for Week 12 Days 78-84 were used (Day 1 corresponds to start of treatment). These data were aggregated to a mean daily frequency as (total number of moderate to severe HF during that week) / (total number of available days with data during that week). In case data is not available for more than 2 days within a week, the value for that particular week was be set to missing.
Time Frame: From baseline to Week 30
Population: FAS
Measure: Mean (Standard Deviation); unit: Hot flashes per day
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Hot flashes per day
  Baseline: number analyzed (Participants) | 199 | 200
  Baseline | 14.66 (11.08) | 16.16 (11.15)
  Change from baseline to Week 1: number analyzed (Participants) | 198 | 197
  Change from baseline to Week 1 | -4.66 (6.70) | -3.57 (6.86)
  Change from baseline to Week 4: number analyzed (Participants) | 185 | 192
  Change from baseline to Week 4 | -8.58 (9.16) | -6.07 (8.91)
  Change from baseline to Week 8: number analyzed (Participants) | 178 | 181
  Change from baseline to Week 8 | -9.67 (10.02) | -6.91 (9.07)
  Change from baseline to Week 12: number analyzed (Participants) | 174 | 180
  Change from baseline to Week 12 | -9.96 (10.25) | -7.24 (8.49)
  Change from baseline to Week 16: number analyzed (Participants) | 166 | 175
  Change from baseline to Week 16 | -10.96 (11.55) | -10.89 (9.54)
  Change from baseline to Week 20: number analyzed (Participants) | 162 | 169
  Change from baseline to Week 20 | -11.60 (11.54) | -11.26 (9.31)
  Change from baseline to Week 26: number analyzed (Participants) | 108 | 120
  Change from baseline to Week 26 | -11.76 (11.38) | -12.76 (12.28)
  Change from baseline to Week 30: number analyzed (Participants) | 132 | 134
  Change from baseline to Week 30 | -7.90 (11.68) | -9.36 (11.71)

7. Secondary Outcome: Mean Change in Patient-reported Outcomes Measurement Information System Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) Total T-score From Baseline to Week 12
Description: In controversy of what you have been proposing above here you are just explaining the PROMIS SD SF 8b scores, not the secondary endpoint which is the change in the T-scores from BL to week 12
  The PROMIS Sleep Disturbance Short Form 8b (PROMIS SD SF 8b) measures sleep disturbance over the past 7 days using 8 items assessing sleep quality, depth, restorative sleep, difficulty falling or staying asleep, and perceptions of sleep adequacy and satisfaction. Items use 5-point response options that vary by item (e.g., Not at all → Very much; Never → Always; Very poor → Very good). Item scores sum to a raw score of 8-40, which is converted to a T-score (mean 50, SD 10; range 28.9-76.5). Higher scores reflect greater sleep disturbance. PROMIS cut points classify T-scores of 55-59 as mild, 60-69 as moderate, and ≥70 as severe disturbance.
Time Frame: From baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Scores on a scale
  Baseline: number analyzed (Participants) | 188 | 193
  Baseline | 61.7 (6.2) | 60.7 (7.2)
  Change from baseline: number analyzed (Participants) | 161 | 172
  Change from baseline | -10.6 (7.7) | -5.5 (6.9)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p < 0.0001, MMRM — [p-value comment as in outcome 1, analysis 1]; LS-means = -4.32, 95% CI 2-sided [-5.77 to -2.86]

8. Secondary Outcome: Mean Change in Menopause-specific Quality of Life Scale (MENQOL) Total Score From Baseline to Week 12
Description: The MENQOL questionnaire was comprised of 29 items assessing the presence of menopausal symptoms and the impact of menopause on health-related quality of life over the past week. The items assessed four domains of symptoms and functioning: VMS, psychosocial functioning, physical functioning, and sexual functioning. For each item, the participants indicated if they had experienced the symptom (yes/no). If participants selected yes, participants rated how bothered they were by the symptom using a six-point verbal descriptor scale, with response options ranging from 0 'not at all bothered' to 6 'extremely bothered'. Based on the individual responses, item scores, domain scores, and a total MENQOL score were calculated. The four domain scores were calculated as a mean of converted single item scores (range 1-8), and the mean of the four domain scores yielded the MENQOL total score. Higher scores indicated greater bother.
Time Frame: From baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Scores on a scale
  Baseline: number analyzed (Participants) | 186 | 189
  Baseline | 4.48 (1.14) | 4.49 (1.17)
  Change from baseline: number analyzed (Participants) | 157 | 167
  Change from baseline | -1.34 (1.29) | -0.97 (1.16)
Statistical Analysis 1: Comparison: Elinzanetant 120 mg vs Placebo - Elinzanetant 120 mg; Test type: Superiority; p = 0.0059, MMRM — [p-value comment as in outcome 1, analysis 1]; LS-means = -0.30, 95% CI 2-sided [-0.53 to -0.07]

9. Secondary Outcome: Mean Change in Beck Depression Inventory (BDI-II) Total Score From Baseline to Week 12
Description: The BDI-II consisted of 21 items to assess the severity of depression over the past 2 weeks. Each item was a list of four statements arranged in increasing levels of severity about a particular symptom of depression. Items used a 4-point verbal response scale ranging from 0 (not at all) to 3 (extreme form of each symptom); specific response options were tailored to the aspect of depression being measured in each item. A total score ranging from 0 to 63 was calculated with scores of 0-13 indicating mild minimal range, 14 - 19 indicating mild depression, 20 - 28 indicating moderate and 29 - 63 indicating severe depression (higher score = greater depression).
Time Frame: From baseline to Week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Scores on a scale
  Baseline | 6.6 (6.5) | 7.2 (6.8)
  Change from baseline: number analyzed (Participants) | 170 | 174
  Change from baseline | -0.2 (8.3) | 0.8 (8.6)

10. Secondary Outcome: Mean Change in BDI-II Total Score From Baseline to Week 26
Description: as for outcome 9
Time Frame: From baseline to Week 26
Population: FAS
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Elinzanetant 120 mg | Placebo - Elinzanetant 120 mg
Number analyzed (Participants) | 200 | 200
Scores on a scale
  Baseline | 6.6 (6.5) | 7.2 (6.8)
  Change from baseline: number analyzed (Participants) | 111 | 110
  Change from baseline | -1.0 (6.9) | -1.1 (6.7)

ADVERSE EVENTS:
Time Frame: From the start of study medication up to 14 days after the last dose of medication, approximately 28 weeks. Adverse event reporting for the all-cause mortality considers all deaths that occurred at any time during the study before the last contact, approximately 30 weeks.
Groups:
- Elinzanetant 120mg Week 1-12: Participants who received elinzanetant 120 mg during Weeks 1-12. Reported AEs for the exposure period Week 1-12 to elinzanetant.
- Placebo Week 1-12: Participants who received placebo during Weeks 1-12. Reported AEs for the exposure period to placebo.
- Elinzanetant 120mg Week 13-26: Participants who received elinzanetant 120 mg during Week 1-12 and continued with elinzanetant 120 mg after Week 12. Reported AEs for the exposure period Week 13 - 26 to elinzanetant.
- Placebo - Elinzanetant 120mg Week 13-26: Participants who received placebo during Weeks 1-12 and switched to elinzanetant 120 mg after Week 12. Reported AEs for the exposure period to elinzanetant.
- Elinzanetant 120mg Week 1-26: Participants who received elinzanetant 120 mg at any time during the study (including those who switched from placebo to elinzanetant 120 mg at Week 13). Reported AEs for the exposure period to elinzanetant for both treatment groups.
Arm/Group | Elinzanetant 120mg Week 1-12 | Placebo Week 1-12 | Elinzanetant 120mg Week 13-26 | Placebo - Elinzanetant 120mg Week 13-26 | Elinzanetant 120mg Week 1-26
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/199 | 0/171 | 0/180 | 0/381
Serious Adverse Events (participants affected / at risk) | 1/201 | 1/199 | 1/171 | 3/180 | 5/381
Other Adverse Events (participants affected / at risk) | 34/201 | 25/199 | 5/171 | 8/180 | 45/381
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant 120mg Week 1-12 (N=201) | Placebo Week 1-12 (N=199) | Elinzanetant 120mg Week 13-26 (N=171) | Placebo - Elinzanetant 120mg Week 13-26 (N=180) | Elinzanetant 120mg Week 1-26 (N=381)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device loosening (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elinzanetant 120mg Week 1-12 (N=201) | Placebo Week 1-12 (N=199) | Elinzanetant 120mg Week 13-26 (N=171) | Placebo - Elinzanetant 120mg Week 13-26 (N=180) | Elinzanetant 120mg Week 1-26 (N=381)
Fatigue (General disorders) | 11 (14) | 3 (3) | 1 (1) | 3 (3) | 15 (18)
Depression rating scale score increased (Investigations) | 9 (10) | 17 (19) | 0 (0) | 2 (2) | 11 (12)
Headache (Nervous system disorders) | 18 (21) | 5 (5) | 4 (5) | 4 (4) | 24 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI will submit any proposed publications to the sponsor, who may advise PI within 30 days of any information that is confidential or requires protection and may request to remove confidential information or delay the publication for 60 days. For this multicenter study, PI will not, without the sponsor's consent, publish results until a multicenter publication is published; if that is not done within 12 months after study completion, PI may publish results in accordance with above provisions.

DOCUMENTS (2):
  • Study Protocol (2022-06-22): https://cdn.clinicaltrials.gov/large-docs/59/NCT05099159/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT05099159/SAP_001.pdf